CLINICAL TRIAL: NCT02696187
Title: Feasibility and Effects of KOL-webben - an Internet Based Health Promotion Tool Directed Towards People With Chronic Obstructive Pulmonary Disease and Staff in the Primary Health Care in Sweden
Brief Title: Feasibility and Effects of KOL-webben in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KOLwebben
Record Dates: First submitted 2016-01-14; First posted 2016-03-02 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Feasibility; Health promotion tool; Self management; Evidence based care; Knowledge transfer; Implementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KOLwebben (Experimental): Patients in the experimental group will be introduced to KOL-webben during their ordinary visits to the primary care center. All patients will receive a pedometer
  Interventions: Behavioral: KOLwebben
- Control group (No Intervention): Other than receiving a pedometer the patients in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: KOLwebben — KOL-webben will be introduced to all people with COPD during their ordinary visits to the primary care center during a 3 months period. The introduction to KOL-webben will be tailored to each person's needs and include 1) registration of the patient at KOL-webben 2) showing and discussing specific content on KOL-webben (e.g. movies with exercises if the person needs exercise training) chosen to meet the needs of the individual 3) giving a card (A5 format) with address to KOL-webben, user information and references to chosen content on KOL-webben. All patients will also receive a pedometer.
  Arms: KOLwebben

SUMMARY:
This study evaluates the effects of KOL-webben (the COPD web), an interactive web-based system directed towards two target groups; people with chronic obstructive pulmonary disease (COPD) and health professionals in primary care. KOL-webben include tools that improve health literacy with a specific focus on 1) increased physical activity and 2) use of appropriate self-management strategies. Moreover, KOL-webben include knowledge and tools directed towards staff in the primary care aimed to implement provision of evidence based health promotion interventions.The feasibility and effects of KOL-webben will be evaluated.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is a cornerstone in the management of patients with chronic obstructive pulmonary disease (COPD) and includes self-management strategies and exercise training. Pulmonary rehabilitation has been shown to decrease dyspnea, improve physical capacity, level of physical activity and health-related quality of life. Traditionally patients with COPD have been treated at pulmonary or medical departments in hospitals. However, due to changes in the Swedish health system these patients now are mainly treated in primary care. Though, the pulmonary rehabilitation programs are still mainly offered by hospitals.

Our research group performed a survey in all hospitals treating patients with COPD in Sweden. The investigators found that less than a half percent of the COPD population took part in pulmonary rehabilitation in 2011. Moreover, a recent survey study performed in Swedish primary care settings found that physiotherapists were available for patients with COPD which is positive. However, only 10 % of the patients with COPD have had access to physiotherapy for their disease. Consequently there is an urgent need to find new strategies to facilitate the provision of pulmonary rehabilitation in the primary care and to provide to people with COPD.

The components included in pulmonary rehabilitation can be considered as health promotion intervention. Health promotion interventions are an important part of the primary care's assignment/mission in Sweden and in order to stress the responsibility for these interventions directed to people with COPD, we have chosen to use the term health promotion interventions instead of pulmonary rehabilitation. Even though there is strong scientific evidence for beneficial effects of health promoting interventions including physical exercise and self-management strategies, a very limited proportion of the people with COPD get access to such services in the primary care. There is an obvious need to find ways to implement available knowledge in clinical practice. Accordingly, KOL-webben is developed as a method (measure/tool) to implement evidence based health promotion interventions and to facilitate the delivery of such services to people with COPD. KOL-webben is also developed as a tool that will support self-management including health promotion among people with COPD.

The design of the explorative feasibility study will be an controlled study with a baseline assessment, delivery of the intervention during 3 months and a follow-up at two month after the completion of the delivery. In order to explore best practice, the usefulness and the effect of the intervention, the feasibility of the data collection and recruitment of people with COPD, a process evaluation will be carried out.Two primary health care units in the county council of Västerbotten in northern Sweden and four primary units in the county council of Dalarna in Mid Sweden will be included in the study. The units will represent both rural and urban settings.

KOL-webben is an interactive web-based system directed towards two target groups; people with COPD and health care professionals. The section directed towards people with COPD will provide tools that improve health literacy and thereby promote and enable a healthier lifestyle with a specific focus on 1) increased physical activity and 2) use appropriate self-management strategies. The tools include educational material, use of (e.g. texts, images, movies, web-links) and interactive components (e.g. ability to report steps per day and symptoms with feedback) adapted to the different stages of the disease. The section directed towards health care professionals includes tools that aim to improve the knowledge, attitudes and confidence in providing evidence based health promotion interventions. The tools include easily accessible knowledge and material (e.g. movies, screening tests, images, power point presentation for patient education and exercise programs).The control group will be recruited from the same health care units among listed patients with no planned visit within the 3 month intervention period. The control group will not receive any intervention.

* All persons with COPD who visits the primary care centre during the study period will constitute the sample in the intervention group (KOL-webben).
* The control group will be recruited from the same primary health care units among listed patients with no planned visit within the 3 month intervention period
* A subgroup of 40 persons (8 from each unit) will be included in additional assessment according to the following: measure of physical activity, measure of physical activity and the process evaluation, or the process evaluation alone. The subgroup will be consecutively recruited among those who visit the primary care centres. Measures of physical activity will also be made in a similar size subgroup of participants in the control group.

Before and after the three month intervention period effects on impact of COPD in daily life, health literacy, confidence in managing their COPD, aspects of physical activity, self-efficacy to perform physical activity, quality of life, dyspnea and level of physical activity will be collected. In addition will we determine effects on instrumental and conceptual knowledge among health professionals

ELIGIBILITY:
Inclusion Criteria:

* Adults 40 years and above diagnosed with COPD according to GOLD criteria i.e. Forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) < 0.70.
* Needs to understand Swedish or have access to anyone who understands Swedish.

Exclusion Criteria:

* Not COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change in impact of COPD in daily life | Baseline and 3 months after baseline
  Impact of COPD in daily life will be assessed using the COPD assessment test.

SECONDARY OUTCOMES:
Change in health literacy | Baseline and 3 months after baseline
  Health literacy will be assessed using the Swedish C & C HL Scale.
Change in confidence in managing their COPD | Baseline and 3 months after baseline
  Confidence in managing their COPD will be assessed using questions specifically developed for this study (face validity will be tested)
Change in aspects of physical activity | Baseline and 3 months after baseline
  Aspects of physical activity will be assessed using the Grimby's Activity Scale
Change in aspects of physical activity | Baseline and 3 months after baseline
  Aspects of physical activity will be assessed using indicators about physical activity retrieved from the National Board of Health and Welfare
Change in self-efficacy to perform physical activity | Baseline and 3 months after baseline
  Self-efficacy to perform physical activity will be assessed using The SCI Exercise Self-Efficacy Scale (ESES).
Change in quality of life | Baseline and 3 months after baseline
  Quality of life will be assessed using the EQ5D.
Change in dyspnea severity | Baseline and 3 months after baseline
  Dyspnea severity will be assessed using the Medical Research Council Scale.
Change in level of physical activity | 7 Days at baseline and and 7 days at 3 months after baseline
  Level of physical activity will be measured with an activity monitor, the DynaPort MiniMod. The activity monitor data collected during 7 Days at baseline and 7 Days 3 months after baseline will be used to assess change in level of physical activity.
Change in instrumental knowledge among health professionals | Baseline and 3 months after baseline
  Instrumental knowledge use of evidence based health promotion interventions will be assessed through a review of medical records; a baseline review of medical record of patients with a COPD diagnosis who have visited the primary care centre during August and September 2015 will be performed and a follow-up review will be performed after the end of the study period.
Change in conceptual knowledge among health professionals | Baseline and 3 months after baseline
  Conceptual knowledge use (i.e. knowledge, attitudes, and intentions) will be assessed using a questionnaire including both structured and semi-structured questions at baseline and at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wadell, PhD, Principal Investigator — Umeå University; Andre Nyberg, PhD, Study Director — Umeå University; Malin Tistad, PhD, Study Director — Umeå University
Locations (1):
- Umeå university, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyberg A, Sondell A, Lundell S, Marklund S, Tistad M, Wadell K. Experiences of Using an Electronic Health Tool Among Health Care Professionals Involved in Chronic Obstructive Pulmonary Disease Management: Qualitative Analysis. JMIR Hum Factors. 2023 Mar 30;10:e43269. doi: 10.2196/43269. PMID 36995743
- [Derived] Marklund S, Tistad M, Lundell S, Ostrand L, Sorlin A, Bostrom C, Wadell K, Nyberg A. Experiences and Factors Affecting Usage of an eHealth Tool for Self-Management Among People With Chronic Obstructive Pulmonary Disease: Qualitative Study. J Med Internet Res. 2021 Apr 30;23(4):e25672. doi: 10.2196/25672. PMID 33929327
- [Derived] Nyberg A, Wadell K, Lindgren H, Tistad M. Internet-based support for self-management strategies for people with COPD-protocol for a controlled pragmatic pilot trial of effectiveness and a process evaluation in primary healthcare. BMJ Open. 2017 Aug 1;7(7):e016851. doi: 10.1136/bmjopen-2017-016851. PMID 28765136